CLINICAL TRIAL: NCT06539312
Title: Project ASTHMA - Aligning With Schools To Help Manage Asthma and Decrease Health Inequities
Brief Title: Project ASTHMA - Aligning With Schools To Help Manage Asthma and Improve Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Lucy Holmes, MD, Clinical Associate Professor of Pediatrics, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00007712; R01MD018384 (NIH)
Record Dates: First submitted 2024-07-31; First posted 2024-08-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-04

CONDITIONS: Asthma in Children; Directly Observed Therapy
Keywords: Asthma; Children; School-based health center; NIH Guideline-based care; Controller medication; Directly Observed Therapy
MeSH Terms: conditions — Directly Observed Therapy; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBHC group (Experimental)
  Interventions: Other: APP assessment and management of asthma
- PCP group (No Intervention)

INTERVENTIONS:
Other: APP assessment and management of asthma — APPs will be trained to follow NIH guidelines for assessment and management of asthma, and to apply their knowledge to the care of the students. Students will also receive DOT of the morning dose of their controller medication.
  Other Names: DOT of morning dose of controller medication
  Arms: SBHC group

SUMMARY:
Children with asthma from communities that experience health inequities frequently do not receive guideline-based asthma care, and as a result, account for a disproportionate percentage of asthma exacerbations, emergency department visits, and hospitalizations. Project ASTHMA (Aligning with Schools To Help Manage Asthma) tests the effectiveness of school-based health centers as a delivery model to improve health outcomes by providing children with guideline-based asthma assessments and preventive medication management, directly observed therapy of their preventive medication to support adherence, and self-management support. If successful, this multicomponent intervention will represent a cost effective and sustainable model to reduce asthma morbidity in historically marginalized communities, and has the potential to impact communities throughout the United States where over 2,500 school-based health centers operate.

ELIGIBILITY:
Inclusion Criteria:

* uncontrolled asthma

Exclusion Criteria:

* other chronic lung disease such as cystic fibrosis

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Asthma exacerbations | from 1 month after enrollment to the end of the school year for 1 school year; to be assessed after the end of the school year.
  Number of asthma exacerbations requiring systemic steroids based on medical records

SECONDARY OUTCOMES:
Daytime asthma symptoms | to be assessed at baseline and 1-, 3-, 5- and 7-months after enrollment for 1 school year
  Frequency of daytime asthma symptoms based on questionnaire minimum value: 0 days maximum value: 28 days Higher scores mean a worse outcome.
Nighttime asthma symptoms | to be assessed at baseline and 1-, 3-, 5- and 7-months after enrollment for 1 school year
  Frequency of nighttime asthma symptoms based on questionnaire minimum value: 0 nights maximum value: 28 nights Higher scores mean a worse outcome.
Spirometry - FEV1 | to be assessed at baseline and 1-, 3-, 5- and 7-months after enrollment for 1 school year
  Forced Expiratory Volume in 1 second
Spirometry - FEV1/FVC ratio | to be assessed at baseline and 1-, 3-, 5- and 7-months after enrollment for 1 school year
  FEV1/Forced Vital Capacity ratio
ED visits | from 1 month after enrollment to the end of the school year for 1 school year; to be assessed after the end of the school year.
  Number of ED visits for asthma symptoms based on medical records
Urgent care visits | from 1 month after enrollment to the end of the school year for 1 school year; to be assessed after the end of the school year.
  Number of urgent care visits for asthma symptoms based on medical records
Hospitalizations | from 1 month after enrollment to the end of the school year; to be assessed after the end of the school year.
  Number of hospitalizations based on medical records
Quality of Life - caregiver | to be assessed at baseline and at 7-month follow-up for 1 school year
  Children's Health Survey for Asthma, American Academy of Pediatrics Higher scores mean a better outcome.
Activity Limitation | to be assessed at baseline and 1-, 3-, 5- and 7-months after enrollment for 1 school year
  Degree of activity limitation based on questionnaire Higher scores mean a worse outcome.
school absenteeism | from 1 month after enrollment to the end of the school year for 1 school year; to be assessed after the end of the school year.
  Number of missed school days based on school records

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Department of Pediatrics, Buffalo, New York, United States